CLINICAL TRIAL: NCT01502709
Title: Randomized Blinded Placebo-Controlled Clinical Trial of Caloric Vestibular Neurostimulation in Patients With Chronic TMD
Brief Title: Neurostimulation in Temporomandibular Disorders (TMD) Patients
Acronym: CVS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruiting difficulties
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Asma Khan, BDS, PhD, Assistant Professor UNC School of Dentistry, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVS-TMD-001
Record Dates: First submitted 2011-12-06; First posted 2012-01-02 (Estimated); Results first posted 2016-04-26 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Single blind; Randomized; Controlled clinical trial
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caloric Vestibular Neurostimulation (Experimental): Subjects received caloric vestibular neurostimulation
  Interventions: Device: Caloric Vestibular Neurostimulation
- Placebo Arm (Placebo Comparator): Subjects received placebo
  Interventions: Device: placebo

INTERVENTIONS:
Device: Caloric Vestibular Neurostimulation — 1 treatments of caloric vestibular neurostimulation for 7.5 minutes in the right ear
  Arms: Caloric Vestibular Neurostimulation
Device: placebo — Matching placebo device
  Arms: Placebo Arm

SUMMARY:
The investigators propose to conduct a randomized blinded placebo-controlled clinical trial in patients with chronic TMD (N=20). Patients will be randomly assigned to receive either active treatment (caloric vestibular neurostimulation) or placebo. Data will be collected prior to and after treatment on thermal and mechanical pain thresholds, clinical signs and symptoms of TMD, and any adverse events.

DETAILED DESCRIPTION:
Temporomandibular disorders (TMD) are musculoskeletal pain conditions characterized by pain in the temporomandibular joint and/or the masticatory muscles. TMD are amongst the most common chronic musculoskeletal conditions affecting 6 to 12% of the general population yet there are no medicines approved specifically for its treatment. TMD cause substantial suffering and TMD pain is the most common symptom that compels patients to seek therapy. One study found average ratings of pain intensity due to TMD of 4.3 on a 10-point scale, similar to the averages reported for chest pain and back pain. Studies consistently find that TMD has a pronounced impact on quality of life. Thus, a new successful approach to TMD therapy would have a significant clinical and economic impact.

Caloric vestibular stimulation (CVS) is a routine diagnostic test for the assessment of vestibular function and Central nervous system pathology. It is usually conducted by instilling cold or warm water into the external ear canal and has been shown to activate anterior cingulate, temporoparietal and insular cortices. In addition to its use as a diagnostic test, CVS has also been shown to reduce pain in several chronic conditions including migraine, phantom limb pain, spinal cord injury, thalamic pain, and complex regional pain syndrome.

Central sensitization is a common feature of the pain conditions shown to be alleviated by CVS. It is a dysfunctional state of the central nervous system in which pain is no longer coupled to a noxious peripheral stimulus. In the presence of central sensitization the response to a noxious stimulus is exaggerated and prolonged (hyperalgesia) and may involve areas outside the site of injury (secondary hyperalgesia). Pain can also arise spontaneously and can be elicited by innocuous stimuli (allodynia). While the neural mechanisms underlying the development of TMD are poorly understood, there is accumulating evidence that central sensitization plays a critical role in TMD pathogenesis. It has been proposed that there is a cyclical process in which TMD pain results in central sensitization that in turn predisposes patients to more pain. Thus any treatment that reverses central sensitization should in turn result in a decrease in pain.

Caloric vestibular stimulation (CVS) is a safe and effective procedure used for the diagnosis of brainstem injury and for balance assessment. As noted already, there have been intriguing observations in the literature suggesting that caloric vestibular stimulation can lead to the abatement of pain. When a caloric stimulation (warm or cool relative to body temperature) is applied to the ear canal, conduction (primarily via dense bone) to the inner ear, and in particular the prominence of the lateral semicircular canal (SCC), sets up convection currents in the endolymph. The resultant deformation of the cupula (membrane spanning the ampula of the SCC) leads to a phasic change in the tonic firing rate of hair cells at the base of the cupula, thereby altering the firing rate of the afferents of the vestibular nerve (thus a device delivering CVS may be viewed as a class of neurostimulator). The afferents map to nuclei in the brainstem (as well as some phylogenetically ancient, direct connections, e.g. to the thalamus and hippocampus) and then to the fastigial nuclei in the cerebellum. It is hypothesized that the method of action of CVS on pain relates to alteration of the phasic firing rate in the vestibular nerve afferents, which in turn alters the activation of the receiving areas (brainstem and cerebellum).

The primary impediment to therapeutic applications of CVS has been the lack of a clinical device that provides controlled, prolonged, and repeatable caloric stimulation. The use of "ice water" irrigation using syringes or even the water/air irrigators used in balance studies are not practical for treatment regimens that extend up to 10 minutes. Further, the applicants believe that a controlled, time-varying thermal waveform is essential to avoid the effects of adaptation of the cupula, which then attenuates control of the phasic firing rate of the hair cells.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* English speaking
* Females with chronic TMD

Exclusion Criteria:

* History of any of the following: Terminal, progressive and /or unstable medical illness; Previous head or neck surgery for neoplasm; current chemotherapy or radiation therapy; facial trauma or orofacial surgery within the last 6 weeks; seizures, history of drug or alcohol abuse; Otologic disorders including chronic vertigo, chronic tinnitus, otitis external, otitis media, mastoiditis and tympanic membrane perforation; Stroke, transient ischemia attacks or Arnold- Chiari malformation; significant cardiac or respiratory disease; epilepsy or neurological disorders such as dementia, brain injury, and brain tumor
* Subjects who score ≥ 31 on the Becks depression inventory (performed at first appointment)
* History of or current destructive nerve therapies, defibrillator, pacemakers, deep brain stimulator, or Implantable nerve stimulators
* Utilization of other alternative or complementary therapies during the study period
* Participation in a clinical trial involving the use of a clinical devise in the last 30 days
* Women who are currently pregnant or nursing.
* Patients who are left handed.
* Current orthodontic treatment.
* Use of an opiate in the 48 hour period preceding the baseline study visit
* The use of anti-histamines 6 hours before, during or immediately after the treatment period
* The use of anti-nausea or anti-vertigo drugs 6 hours before or during the treatment period

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asma Khan, BDS, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill School of Dentistry, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Caloric Vestibular Neurostimulation: 1 treatment of caloric vestibular neurostimulation for 7.5 minutes in the right ear
- Placebo Arm: 0 participants received placebo
Period: Overall Study
Arm/Group | Caloric Vestibular Neurostimulation | Placebo Arm
Started | 5 | 0
Completed | 1 | 0
Not Completed | 4 | 0
Not completed — Lost to Follow-up | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caloric Vestibular Neurostimulation | Placebo Arm | Total
Number analyzed (Participants) | 5 | 0 | 5
Age, Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 5 |  | 5
  >=65 years | 0 |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (10.8) |  | 48 (10.8)
Gender [Number; unit: participants]
  Female | 5 |  | 5
  Male | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 |  | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Visual Analog Score (VAS) in Days 1-7 Post Treatment
Description: The mean of measures taken from days 1-7 was calculated. Pain was assessed by using VAS score ranges from 0 millimeter (mm) = no pain to 100 mm = worst possible pain. A decrease in score from Baseline represented treatment response.
Time Frame: Daily Self-reports at Baseline and on Days 1 through 7
Measure: Mean (Standard Deviation); unit: millimeters
Groups:
- Neurostimulator: 1 treatments of caloric vestibular neurostimulation for 7.5 minutes in the right ear
Arm/Group | Neurostimulator | Placebo Arm
Number analyzed (Participants) | 1 | 0
millimeters | 30 (NA) — Data not analyzed because only complete information for 1 subject was available. |

2. Secondary Outcome: Mean Percentage of Time Spent in Pain From Days 1-7
Description: The mean of measures taken from days 1-7 was calculated. Composite pain is a measure of mean pain intensity experienced and pain duration. Pain was assessed by using VAS score ranges from 0 millimeter (mm) = no pain to 100 mm = worst possible pain. Duration of pain ranges from 0 to 100% of a day. For example a pain free subject would report O pain intensity for 0% of the day.
Time Frame: Days 1-7
Measure: Mean (Standard Deviation); unit: percentage of day in pain
Arm/Group | Caloric Vestibular Neurostimulation | Placebo Arm
Number analyzed (Participants) | 1 | 0
percentage of day in pain | 77 (NA) — Data not analyzed because only complete information for 1 subject was available. |

3. Secondary Outcome: Number of Participants With Signs and Symptoms of Temporomandibular Disorder Based on Outcomes of Research Diagnostic Criteria (RDC) Exam
Description: RDC for Temporomandibular disorders (TMD) is a reliable & valid system for diagnosis of TMD, utilizing clinical procedures, diagnostic algorithms, and a dual-axis assessment comprising symptom history and physical exam. Signs and symptoms were evaluated by a trained professional and the history was obtained through use of questionnaires. In all sections and scales the higher the number reported corresponds to the more pain being experienced, therefore, a worse outcome. The clinical exam consists of facial, dental, and cervical evaluations including mandibular range of motion, Temporomandibular disorders Joint sound, and palpation of the orofacial muscles and temporomandibular joints (TMJ). Subjects are classified as TMD if they report pain in or around the temporomandibular joints or muscles of mastication for more than 3 months.
Time Frame: Baseline, Month 3
Measure: Number; unit: Participants
Arm/Group | Caloric Vestibular Neurostimulation | Placebo Arm
Number analyzed (Participants) | 1 | 0
Participants | 1 |

ADVERSE EVENTS:
Time Frame: 2 hours post-treatment
Arm/Group | Caloric Vestibular Neurostimulation | Placebo Arm
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/0
Other Adverse Events (participants affected / at risk) | 4/5 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caloric Vestibular Neurostimulation (N=5) | Placebo Arm (N=0)
Facial flushing (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Mild, transient
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dry Mouth (General disorders) | 3 (3) | 0 (0)
Feeling Cold (General disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No